CLINICAL TRIAL: NCT04346368
Title: Safety and Efficacy of Intravenous Infusion of Bone Marrow-Derived Mesenchymal Stem Cells in Severe Patients With Coronavirus Disease 2019 (COVID-19): A Phase 1/2 Randomized Controlled Trial
Brief Title: Bone Marrow-Derived Mesenchymal Stem Cell Treatment for Severe Patients With Coronavirus Disease 2019 (COVID-19)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Collaborators: Guangzhou Eighth People's Hospital (Unknown); Tongji Hospital (Other); Guangzhou Cellgenes Biotechnology Co.,Ltd (Unknown)
Responsible Party: Principal Investigator, ShiYue Li, Professor, Guangzhou Institute of Respiratory Disease
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SC-2020-01
Record Dates: First submitted 2020-03-23; First posted 2020-04-15 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Coronavirus Disease 2019 (COVID-19)
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bone Marrow-Derived Mesenchymal Stem Cells (BM-MSCs) (Experimental): Conventional treatment plus BM-MSCs
  Interventions: Biological: BM-MSCs
- Placebo (Placebo Comparator): Conventional treatment plus placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: BM-MSCs — Participants will receive conventional treatment plus BM-MSCs(1*10E6 /kg body weight intravenously at Day 1).
  Arms: Bone Marrow-Derived Mesenchymal Stem Cells (BM-MSCs)
Biological: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Coronavirus Disease 2019 (COVID-19) is spreading worldwide and has become a public health emergency of major international concern. Currently, no specific drugs or vaccines are available. For severe cases, it was found that aberrant pathogenic T cells and inflammatory monocytes are rapidly activated and then producing a large number of cytokines and inducing an inflammatory storm.Mesenchymal stem cells (MSCs) have been shown to possess a comprehensive powerful immunomodulatory function. This study aims to investigate the safety and efficacy of intravenous infusion of mesenchymal stem cells in severe patients with COVID-19.

DETAILED DESCRIPTION:
COVID-19 has become a urgent and serious public health event that threatens human life and health globally. No specific pharmacological treatments are available to date for COVID-19.Patients contracting the severe form of the disease constitute approximately 15% of the cases which is characterized by extensive acute inflammation. In these severe cases, there will be rapid respiratory system failure.

MSCs have been employed extensively in cell therapy, which includes a plethora of preclinical research investigations as well as a significant number of clinical trials. Safety and efficacy have been shown in many clinical trials. Previous studies have shown that MSCs could significantly reduce inflammatory cell infiltration in lung tissue, reduce inflammation in lung tissue, and significantly improve lung The structure and function of tissues protect lung tissue from damage.The mechanisms underlying the improvements after MSC infusion in COVID-19 patients also appeared to be the robust antiinflammatory activity of MSCs. Recent studies also showed that intravenous MSC infusion could reduce the overactivation of the immune system and support repair by modulating the lung microenvironment after SARS-CoV-2 infection. MSC therapy inhibiting the overactivation of the immune system and promoting endogenous repair by improving the lung microenvironment after the SARS-CoV-2 infection.

The purpose of this study is to investigate the safety and efficacy of intravenous infusion of mesenchymal stem cells in severe patients With COVID-19.The respiratory function, pulmonary inflammation, clinical symptoms, pulmonary imaging, side effects, immunological characteristics will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent prior to performing study procedures
2. Age ≥18 years, and ≤75 years;

   A confirmed case of Covid-19. The criteria are as follows:

   Clinically diagnosed or suspected cases with one of the following etiological evidence: 1) SARS-CoV-2 nucleic acid is positive in respiratory or blood samples detected by RT-PCR; 2) virus sequence detected in respiratory or blood samples shares high homology with the known sequence of SARS-CoV-2.
3. Clinical classification is severe case: Meet any of the following:

1) Increased respiratory rate (≥30 beats / min), difficulty breathing, cyanosis of the lips; 2) Peripheral capillary oxygen saturation (SpO2) ≤93% at rest ; 3)Partial pressure of arterial oxygen (PaO2) / Fraction of inspired oxygen (FiO2) ≤300 mmHg (1mmHg = 0.133kPa).

Exclusion Criteria:

1. Other types of viral pneumonia, or bacterial pneumonia.
2. The clinical classification is mild, moderate or critical;
3. Patients with malignant blood or solid tumor.
4. Pregnant or lactating women;
5. There are other situations or diseases that the investigator think are not suitable to participate in this clinical study or may be increased risk of the subject.
6. Patients with serious social and mental disability, inability/restriction of legal capacity;
7. Refusal to sign informed consent;
8. Patients with severe liver disease (eg Child Pugh score ≥ C, AST> 5 times upper limit of normal );
9. Patients with severe renal insufficiency (estimated glomerular filtration rate ≤30mL / min / 1.73m2) or receiving continuous renal replacement therapy, hemodialysis, peritoneal dialysis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Changes of oxygenation index (PaO2/FiO2) | At baseline, 6 hour, Day 1, Day 3,Week 1, Week 2, Week 4, Month 6.
  Evaluation of pneumonia improvement
Side effects in the BM-MSCs treatment group | Baseline through 6 months
  Proportion of participants with treatment-related adverse events

SECONDARY OUTCOMES:
Clinical outcome | At baseline, 6 hour, Day 1, Day 3,Week 1, Week 2, Week 4, Month 6.
  Improvement of clinical symptoms including duration of fever, respiratory destress, pneumonia, cough, sneezing, diarrhea.
Hospital stay | Baseline through 6 months
  days of the patients in hospital
CT Scan | At baseline, 6 hour, Day 1, Day 3,Week 1, Week 2, Week 4, Month 6.
  Evaluation of pneumonia improvement
Changes in viral load | At baseline, 6 hour, Day 1, Day 3,Week 1, Week 2, Week 4, Month 6.
  (deep sputum / pharyngeal swab / nasal swab / anal swab / tear fluid / stomach fluid / feces / blood or alveolar lavage fluid)
Changes of CD4+, CD8+ cells count and concentration of cytokines | At baseline, 6 hour, Day 1, Day 3,Week 1, Week 2, Week 4, Month 6.
  Immunological status
Rate of mortality within 28-days | From baseline to day 28
  Marker for efficacy
Changes of C-reactive protein | At baseline, 6 hour, Day 1, Day 3,Week 1, Week 2, Week 4, Month 6.
  Markers of Infection

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Institute of Respiratory Health, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China